CLINICAL TRIAL: NCT00982657
Title: A Phase Ib/ii, Multicenter, Trial Of Cvx-060, A Selective Angiopoietin-2 (Ang-2) Binding, Anti-angiogenic Covx-body, In Combination With Sunitinib In Patients With Advanced Renal Cell Carcinoma
Brief Title: A Trial Of CVX-060, An Anti-Angiogenic COVX-Body, In Combination With Sunitinib In Patients With Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Refer to statement in Summary Section/Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1131001; CVX-060-102 (Other: Alias Study Number); 2010-022657-42 (EudraCT Number)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Solid Tumor
Keywords: Phase Ib Phase II Advanced solid tumor Clear cell renal cancer Sunitinib plus / minus CVX-060
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): CVX-060 + sunitinib
  Interventions: Drug: CVX-060 + sunitinib
- Cohort 2 (Experimental): CVX-060 + sunitinib
  Interventions: Drug: CVX-060 + sunitinib
- Cohort 3 (Experimental): CVX-060 + sunitinib
  Interventions: Drug: CVX-060 + sunitinib
- Expanded cohort (Experimental): CVX-060 + sunitinib
  Interventions: Drug: CVX-060 + sunitinib
- Phase II - Arm A (Experimental): CVX-060 + sunitinib
  Interventions: Drug: CVX-060 + sunitinib
- Phase II - Arm B (Active Comparator): sunitinib alone
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: CVX-060 + sunitinib — CVX-060 weekly infusions at 6.0 mg/kg + 50 mg sunitinib daily (4 out of 6 weeks)
  Other Names: CVX-060 / Sutent
  Arms: Cohort 1
Drug: CVX-060 + sunitinib — CVX-060 weekly infusions at 12.0 mg/kg + 50 mg sunitinib daily (4 out of 6 weeks)
  Other Names: CVX-060 / Sutent
  Arms: Cohort 2
Drug: CVX-060 + sunitinib — CVX-060 weekly infusions at 15.0 mg/kg + 50 mg sunitinib daily (4 out of 6 weeks)
  Other Names: CVX-060 / Sutent
  Arms: Cohort 3
Drug: CVX-060 + sunitinib — CVX-060 weekly infusions at TBD mg/kg + 50 mg sunitinib daily (4 out of 6 weeks)
  Other Names: CVX-060 / Sutent
  Arms: Expanded cohort
Drug: CVX-060 + sunitinib — CVX-060 weekly infusions at TBD mg/kg + 50 mg sunitinib daily (4 out of 6 weeks)
  Other Names: CVX-060 / Sutent
  Arms: Phase II - Arm A
Drug: Sunitinib — 50 mg sunitinib daily (4 out of 6 weeks)
  Other Names: Sutent
  Arms: Phase II - Arm B

SUMMARY:
The safety and tolerability of CVX-060 have been established in the first-in-human clinical trial, CVX-060-101. Thus, this phase Ib/II trial is to assess the safety and pharmacokinetics (PK) profiles of combining CVX-060 with sunitinib in patients with advanced solid tumors, and to subsequently assess the treatment efficacy of the combination treatment, as well as that of sunitinib alone in patients with advanced renal cell carcinoma (mRCC).

DETAILED DESCRIPTION:
On 23-Nov-2010, B1131001 (CVX-060-102) was closed to enrollment due to emerging clinical data which led to a re-assessment of the strategic goals of the PF-04856884 program. The study enrolled the Phase 1b portion only. Subsequently, on 25-Oct-2012, due to data safety signals in a separate clinical trial with PF-04856884 (CVX-060), all PF-04856884 studies were discontinued and ongoing patients on B1131001 were permitted to remain on study at a reduced PF-04856884 dose if determined to have been deriving clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced/metastatic solid tumor
* Having received at least 1 prior systemic therapy for the treatment of advanced/metastatic solid tumors
* Histologically or cytologically confirmed renal cell carcinoma with clear cell histology and evidence of metastasis (No previous systemic therapy for the treatment of metastatic renal cell carcinoma)
* Adequate laboratory tests
* Eastern Cooperative Oncology Group (ECOG) 0-1, Life expectancy > or = 12 weeks and age > or = 18 years

Exclusion Criteria:

* Patients intolerant of prior anti-angiogenic agents
* Recent history of bleeding or bleeding disorders
* History of tumors in the brain
* History of heart problems
* History of severe allergic reaction to antibody therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Premiere Oncology, A Medical Corporation, Santa Monica, California
  - Boston Baskin Cancer Foundation, Southaven, Mississippi
  - Providence Portland Medical Center, Portland, Oregon
  - Boston Baskin Cancer Foundation, Bartlett, Tennessee
  - Boston Baskin Cancer Foundation, Germantown, Tennessee
  - Boston Baskin Cancer Foundation, Memphis, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1131001&StudyName=A%20Trial%20Of%20CVX-060%2C%20An%20Anti-Angiogenic%20COVX-Body%2C%20In%20Combination%20With%20Sunitinib%20In%20Patients%20With%20Advanced%20Renal%20Cell%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 phases, Phase 1b and Phase 2. On 23 Nov 2010, this study was closed to enrollment due to emerging clinical data which led to a re-assessment of strategic goals of the CVX-060 program. The study enrolled the Phase 1b portion only.
Groups:
- CVX-060 6 mg/kg + Sunitinib 50 mg: CVX-060 6 milligram per kilogram (mg/kg) of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks of off treatment (6-week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
- CVX-060 6 mg/kg + Sunitinib 37.5 mg: CVX-060 6 mg/kg of body weight intravenous infusion administered once-weekly with oral 37.5 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off (6-week cycle) treatment until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
- CVX-060 12 mg/kg + Sunitinib 50 mg: CVX-060 12 mg/kg of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6-week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
- CVX-060 15 mg/kg + Sunitinib 50 mg: CVX-060 15 mg/kg of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6-week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
Period: Overall Study
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Started | 12 | 3 | 3 | 16
Completed | 11 | 3 | 1 | 7
Not Completed | 1 | 0 | 2 | 9
Not completed — Death | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3
Not completed — Other | 0 | 0 | 0 | 4
Not completed — On going at date of cut-off | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis set consisted of all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg | Total
Number analyzed (Participants) | 12 | 3 | 3 | 16 | 34
Age, Customized [Number; unit: Participants]
  Less than (<) 18 years | 0 (9.6) | 0 (8.5) | 0 (8.5) | 0 (13.7) | 0
  18 to 44 years | 0 | 0 | 0 | 2 | 2
  45 to 64 years | 6 | 2 | 3 | 9 | 20
  Greater than or equal to (>=) 65 years | 6 | 1 | 0 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 2 | 4 | 14
  Male | 6 | 1 | 1 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the dose level at which less than or equal to (<=) 1/6 participants experienced Dose Limiting Toxicity (DLT) during the first cycle of treatment with the next higher dose having >= 2/6 participants with DLT.
Time Frame: Baseline up to Cycle 1( Day 1 to Day 42)
Population: The study was terminated during the Phase 1b phase by the sponsor prematurely. Due to the decision of not conducting the Phase II portion of the study, no MTD was assessed.
Groups:
- All Participants: All participants who received 6 mg/kg, 12mg/kg or 15 mg/kg of CVX-060 intravenous infusion along with oral 50 mg or 37.5 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose date to the first documentation of disease progression or death due to any cause, whichever occurred first.
Time Frame: Baseline tumor progression/clinical deterioration or death (up to 28 days post last dose of study medication)
Population: The study was terminated during the Phase 1b phase by the sponsor prematurely. Due to the decision of not conducting the Phase II portion of the study.The PFS endpoint was a pre-specified endpoint for the Phase II portion of the study, and was therefore not assessed.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic Parameters of CVX-060
Description: Pharmacokinetic parameters Area under the Curve (AUC), Maximum Observed Serum Concentration (Cmax), Minimum Observed Serum Trough Concentration (Cmin), Clearance (CL), terminal elimination half life (t1/2) were planned to be analyzed.
Time Frame: Pre-dose on Day 1 Cycle 1 ; post-dose on Day 1, 5, 8, 15, 22, 29 Cycle 1 , Day 1 Cycle 2, to Cycle 28 , end of study (7 days post last dose of study medication), follow-up visit (28 days post last dose of study medication)
Population: The study was terminated during the Phase 1b phase by the sponsor prematurely. Due to the decision of not conducting the phase II portion of the study,pharmacokinetics assessment was not conducted.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: DLT included grade 4 neutropenia of >= 3 day duration or with grade 4 neutropenia associated with fever; grade 4 thrombocytopenia for >= 3 consecutive days; Proteinuria of >=2 grams (g) per 24 hours; inability to resume to CVX-060 or sunitinib within 14 days of scheduled administration due to treatment related toxicity; any Grade 3 nonhematologic toxicity except nausea, vomiting, and diarrhea; Grade 3 nausea, vomiting, or diarrhea which persists for >=48 hours; Any >= Grade 4 non-hematologic toxicity; Any additional hematological or non-hematological toxicity for which dose reduction was required or for which patient was discontinued from the trial.
Time Frame: Baseline up to 28 days post last dose of study medication
Population: Safety Analysis set consisted of all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 12 | 3 | 3 | 16
participants | 2 | 1 | 0 | 2

5. Secondary Outcome: Serum Angiopoietin-2 (Ang-2) and Plasma Vascular Endothelial Growth Factor (VEGF) Levels
Time Frame: Ang-2 (Day 1, 2, 5, 8, 22, 29 Cycle 1, Day 1 Cycle 2 up to Cycle 28); VEGF (Day 1, 8, 15, 22 Cycle 1, Day 1 Cycle 2 up to Cycle 28)
Population: The study was terminated during the Phase 1b phase by the sponsor prematurely. Due to the decision of not conducting the phase II portion of the study, pharmacodynamics assessment was not conducted.
Groups:
- CVX-060 6 mg/kg + Sunitinib 50 mg: CVX-060 6 milligram per kilogram (mg/kg) of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6-week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
- CVX-060 6 mg/kg + Sunitinib 37.5 mg: CVX-060 6 mg/kg of body weight intravenous infusion administered once-weekly with oral 37.5 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6-week cycle) until disease progression, unacceptable toxicity ,withdrawal of consent or investigator's discretion.
- CVX-060 12 mg/kg + Sunitinib 50 mg: CVX-060 12 mg/kg of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6-week cycle) until disease progression, unacceptable toxicity ,withdrawal of consent or investigator's discretion.
- CVX-060 15 mg/kg + Sunitinib 50 mg: CVX-060 15 mg/kg of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6-week cycle) until disease progression, unacceptable toxicity ,withdrawal of consent or investigator's discretion.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs) and Non-Serious Adverse Events (Non-SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre treatment state.
Time Frame: Baseline up to 28 days post last dose of study medication
Population: Safety Analysis set consisted of all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Groups:
- CVX-060 6 mg/kg + Sunitinib 37.5 mg: CVX-060 6 mg/kg of body weight intravenous infusion administered once-weekly with oral 37.5 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6-week cycle) until disease progression, unacceptable toxicity, withdrawal of consent occurred or investigator's discretion.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 12 | 3 | 3 | 16
Participants
  SAEs | 4 | 0 | 1 | 8
  non-SAEs | 12 | 3 | 3 | 16

7. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. Per RECIST v1.0: CR defined as disappearance of all target lesions and non-target lesions. PR defined as >= 30% decrease in sum of the longest diameters (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non target lesions.
Time Frame: Baseline up to 7 days post last dose of study medication
Population: Safety Analysis set consisted of all participants who received at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- CVX-060 6 mg/kg + Sunitinib 50 mg: CVX-060 6 milligram per kilogram (mg/kg) of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6 week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
- CVX-060 6 mg/kg + Sunitinib 37.5 mg: CVX-060 6 mg/kg of body weight intravenous infusion administered once-weekly with oral 37.5 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6 week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
- CVX-060 12 mg/kg + Sunitinib 50 mg: CVX-060 12 mg/kg of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6 week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
- CVX-060 15 mg/kg + Sunitinib 50 mg: CVX-060 15 mg/kg of body weight intravenous infusion administered once-weekly with oral 50 mg sunitinib capsule once daily up to 4 weeks followed by 2 weeks off treatment (6 week cycle) until disease progression, unacceptable toxicity, withdrawal of consent or investigator's discretion.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 12 | 3 | 3 | 12
Percentage of participants | 0 [NA to NA] — Confidence interval (CI) was not estimable because there were no participants with objective response. | 0 [NA to NA] — CI was not estimable because there were no participants with objective response. | 0 [NA to NA] — CI was not estimable because there were no participants with objective response. | 0 [NA to NA] — CI was not estimable because there were no participants with objective response.

8. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or death due to any cause, whichever occurs first. Participants last known to be progression free are censored at the date of the last objective disease assessment that verified lack of disease progression.
Time Frame: Baseline up to 7 days post last dose of study medication
Population: Duration of response was not calculated as there were no participants with objective response.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Anti- CVX-060 Antibodies
Time Frame: Baseline up to 28 days after last CVX-060 dose
Population: The study was terminated during the Phase 1b phase by the sponsor prematurely. Due to the decision of not conducting the phase II portion of the study, no Anti-CVX-060 antibody assessment was conducted.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CVX-060 6 mg/kg + Sunitinib 50 mg | CVX-060 6 mg/kg + Sunitinib 37.5 mg | CVX-060 12 mg/kg + Sunitinib 50 mg | CVX-060 15 mg/kg + Sunitinib 50 mg
Serious Adverse Events (participants affected / at risk) | 4/12 | 0/3 | 1/3 | 8/16
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 3/3 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVX-060 6 mg/kg + Sunitinib 50 mg (N=12) | CVX-060 6 mg/kg + Sunitinib 37.5 mg (N=3) | CVX-060 12 mg/kg + Sunitinib 50 mg (N=3) | CVX-060 15 mg/kg + Sunitinib 50 mg (N=16)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Herpes oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CVX-060 6 mg/kg + Sunitinib 50 mg (N=12) | CVX-060 6 mg/kg + Sunitinib 37.5 mg (N=3) | CVX-060 12 mg/kg + Sunitinib 50 mg (N=3) | CVX-060 15 mg/kg + Sunitinib 50 mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 4
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 1 | 2 | 4
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 1
Periorbital oedema (Eye disorders) | 1 | 0 | 1 | 4
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1
Retinal oedema (Eye disorders) | 0 | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 0 | 0 | 1
Scleral discolouration (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 4
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 2 | 11
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 0 | 1 | 5
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 3
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 2 | 1 | 7
Oesophageal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Tongue geographic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 2 | 8
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2
Chills (General disorders) | 2 | 1 | 0 | 4
Cyst (General disorders) | 1 | 0 | 0 | 0
Early satiety (General disorders) | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 7 | 3 | 2 | 12
Generalised oedema (General disorders) | 1 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 3
Oedema (General disorders) | 2 | 1 | 0 | 0
Oedema peripheral (General disorders) | 5 | 2 | 1 | 3
Pain (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 4
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Occult blood positive (Investigations) | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 4
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 0 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 3
Dysgeusia (Nervous system disorders) | 5 | 0 | 2 | 6
Headache (Nervous system disorders) | 0 | 0 | 0 | 3
Hemisensory neglect (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 3
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 3 | 0 | 1 | 2
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Genital pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Genital swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Facial operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 6 | 1 | 1 | 9

LIMITATIONS AND CAVEATS:
On 25 Oct 2012, due to data safety signals in separate clinical trial with CVX-060, all CVX-060 studies were discontinued. Ongoing participants in B1131001 were permitted to remain on study at a reduced dose if determined to derive clinical benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.